CLINICAL TRIAL: NCT05530746
Title: Study on the Diagnostic Value of Multi-omics Combined Detection for Precancerous Lesions of Colorectal Cancer
Brief Title: Study on the Diagnostic Value of Multi-omics Combined Detection for Precancerous Lesions of CRC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Other Study IDs: multi-omics
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer; Precancerous Lesion; Inflammatory Bowel Diseases
Keywords: multi-omics study; adenoma; Inflammatory Bowel Disease
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Feces and colon histological specimens will be obtained in healthy individuals, patients with non-advanced adenoma, patients with advanced adenomas, patients with Inflammatory bowel disease, and patients with colon cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control: Volunteers with no significant abnormalities on colonoscopy were given informed consent to obtain colon tissue biopsies and fecal specimens.
- Non-advanced adenoma: Patients with non-advanced adenoma were given informed consent to obtain colon tissue biopsies and fecal specimens.
- Advanced adenoma: Patients with advanced adenoma were given informed consent to obtain colon tissue biopsies and fecal specimens.
- Inflammatory bowel disease: Patients with inflammatory bowel disease were given informed consent to obtain colon tissue biopsies and fecal specimens.
- Colorectal cancer: Patients with colorectal cancer were given informed consent to obtain cancer tissue biopsies and fecal specimens.

SUMMARY:
Colorectal cancer (CRC) has become one of the most common malignant tumors in the world, and the key to its prevention and control is early detection and treatment. As colorectal adenoma and inflammatory bowel disease (IBD) are the inevitable precursors of most CRC, screening for colorectal adenoma and IBD is of great importance for preventing CRC. The existing detection methods have high sensitivity for CRC, while limited in colorectal adenoma and IBD. Therefore, exploring a detection method with high sensitivity for colorectal adenoma and IBD is necessary. This project intends to use methylation detection technology, lactic acid modified omics, proteomics, metagenomics, and other omics technology, through the analysis of differences in feces and histological results in healthy volunteers, patients with non-advanced adenoma, patients with advanced adenomas, patients with IBD, and patients with CRC for early screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is between 18-75.
* Patients who have signed informed consent form.

Exclusion Criteria:

* Patients who have undergone colonic resection or polypectomy.
* Patients with abnormal blood coagulation or taking antiplatelets or anticoagulants within 7 days.
* Patients with hereditary colorectal cancer syndrome (including familial adenomatous polyposis).
* Patients with pregnancy, severe chronic cardiopulmonary and renal disease.
* Patients with failed cecal intubation.
* Patients with poor BPQ necessitated a second bowel preparation.
* Patients refusing to participate or to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population was derived from patients at the Gastroenterology Endoscopy Center of Changhai Hospital in Shanghai, China. And the subjects were divided into five groups according to clinical and histopathological characteristics.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Detection of advanced colorectal adenoma | Through study completion, an average of 1 year
  An advanced colorectal adenoma is defined as a colorectal adenoma ≥10 mm, adenoma with tubulovillous or villous histology, or adenoma with high-grade dysplasia

SECONDARY OUTCOMES:
Detection of colorectal cancer | Through study completion, an average of 1 year
  Lesions will be confirmed as malignant by histopathologic examination.
Detection of non-advanced colorectal adenoma | Through study completion, an average of 1 year
  A non-advanced colorectal adenoma is defined as tubular adenoma less than 1cm in diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D, Principal Investigator — Study Principal Investigator
Locations (1):
- Changhai Hospital, Naval Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang D, Tang Z, Huang H, Zhou G, Cui C, Weng Y, Liu W, Kim S, Lee S, Perez-Neut M, Ding J, Czyz D, Hu R, Ye Z, He M, Zheng YG, Shuman HA, Dai L, Ren B, Roeder RG, Becker L, Zhao Y. Metabolic regulation of gene expression by histone lactylation. Nature. 2019 Oct;574(7779):575-580. doi: 10.1038/s41586-019-1678-1. Epub 2019 Oct 23. PMID 31645732
- [Background] Zackular JP, Rogers MA, Ruffin MT 4th, Schloss PD. The human gut microbiome as a screening tool for colorectal cancer. Cancer Prev Res (Phila). 2014 Nov;7(11):1112-21. doi: 10.1158/1940-6207.CAPR-14-0129. Epub 2014 Aug 7. PMID 25104642
- [Background] Wang J, Liu S, Wang H, Zheng L, Zhou C, Li G, Huang R, Wang H, Li C, Fan X, Fu X, Wang X, Guo H, Guan J, Sun Y, Song X, Li Z, Mu D, Sun J, Liu X, Qi Y, Niu F, Chen C, Wu X, Wang X, Song X, Zou H. Robust performance of a novel stool DNA test of methylated SDC2 for colorectal cancer detection: a multicenter clinical study. Clin Epigenetics. 2020 Oct 30;12(1):162. doi: 10.1186/s13148-020-00954-x. PMID 33126908